CLINICAL TRIAL: NCT04936360
Title: Evaluating the Care Burden of Caregivers of Patients With Brain Injury and Determining the Influencing Factors
Status: Completed | Type: Observational
Sponsor: Gaziler Physical Medicine and Rehabilitation Education and Research Hospital (Other)
Responsible Party: Principal Investigator, Yasin Demir, Associate professor, Gaziler Physical Medicine and Rehabilitation Education and Research Hospital
Other Study IDs: 16
Record Dates: First submitted 2021-06-18; First posted 2021-06-23 (Actual); Last update posted 2021-11-29 (Actual); Status verified 2021-05

CONDITIONS: Brain Injuries; Caregiver Burden
Keywords: Caregiver; Brain injury; Burden; Caregiver Strain Index
MeSH Terms: conditions — Brain Injuries; Caregiver Burden | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patient Group: Patients with non-progressive non-neurodegenerative acquired brain damage, who were over 18 years of age, who could establish voluntary social communication will be included in the study.
  Interventions: Other: questionnaires for clinical assessments
- Caregivers Group: Caregivers over the age of 18, who took care of the patient for at least 1 month, and who did not have premorbid medical or psychological problems will be included in the study.
  Interventions: Other: questionnaires for clinical assessments

INTERVENTIONS:
Other: questionnaires for clinical assessments — questionnaires for clinical assessments

SUMMARY:
Acquired brain injury is a general term including trauma due to head injury or postsurgical damage, vascular accident such as stroke or subarachnoid hemorrhage, toxic or metabolic cause such as hypoglycemia, cerebral anoxia, and infection or inflammation. However acquired brain injury leaves survivors with a considerable burden of physical, cognitive, emotional,behavioural and psychosocial limitations,these individuals often require healthcare, supervision, and support from professional or informal caregivers in some or all of their lives. Therefore, this study have two primary aims: (1) to conclude the level of caregiver's life satisfaction and strain; and (2) to determine the factors predicting strain among the caregivers. İnvestigators believe this study can add to the literature and create awareness on the current state of caregiver's well-being in this part of the world.

DETAILED DESCRIPTION:
Patients will evaluate with respect to their demographic and clinical determinants. In the patient group, ambulation status, disability levels, cognitive status, neurobehavioral results, functional status will evaluate with the Functional Ambulation Classification Scale (FACS), Disability Rating Scale (DRS), Rancho Los Amigos Cognitive Scale-Revised (RLAS-R), Neurobehavioral Rating Scale-Revised (NBRS-R), Functional Independence Measure (FIM) respectively. All assessments will conduct and evaluate by the treating physicians during hospitalization.

İnvestigators also will record the type of caregiving (family member or paid professional) and socio-demographic characteristics of the caregivers . Sleep quality will be determined with Pittsburgh Sleep Quality İndex (PSQI), quality of life with NHP (Nottingham Health Profile), level and risk of anxiety and depression with Hospital Anxiety and Depression Scale, satisfaction level with The Satisfaction with Life Scale , care burden with Caregiver Strain Index (CSI).

ELIGIBILITY:
Inclusion criteria for the patients:

* have a nonprogressive, non-neurodegenerative acquired brain injury
* able to read or understand the questionnaire
* at least 18 years of age

Inclusion criteria for the caregivers:

* primary caregiver of a patient diagnosed with acquired brain injury
* at least 18 years of age
* had provided care for at least one month
* providing care to the patient for more than 4 h per day
* did not have any major premorbid medical and psychological illnesses
* able to read or understand the questionnaire

Exclusion criteria for patients and caregivers:

* under 18 years of age
* inability to read and understand questions.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Acquired brain injury patients and their primer caregivers
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2021-04-15 (Actual); Primary Completion 2021-09-15 (Actual); Study Completion 2021-09-15 (Actual)

PRIMARY OUTCOMES:
Functional Independence Measure (FIM) | through study completion, an average of one and a half months
  The FIM measures functional independence with 18 items that assess Self-care (six items), Mobility (seven items), and Cognition (five items). Items are scored 1 through 7 with a score of 1 representing complete dependence and a score of 7 indicating complete independence. The items are summed to obtain a total score ranging from 18 to 126.
Caregiver Strain Index (CSI) | through study completion, an average of one and a half months
  CSI is a 13-item, self-administered objective questionnaire designed to assess level of stress experienced by the informal caregivers. Participants had to answer all the items as either YES or NO. The scoring was one (1) point for each answer of 'YES' and zero (0) for each answer of 'NO'. The question scores were summed with the maximum score of 13. This score was then divided into 'having strain' (score of ≥7) and 'no strain' (score of <7).
The Satisfaction with Life Scale (SWLS) | through study completion, an average of one and a half months
  The SWLS (Satisfaction With Life Scale) provides a global measure of satisfaction with life as an overall summation of a person. It consists of five questions rated on a 7-point Likert scale, from 'strongly agree' (response option 7) to 'strongly disagree' (response option 1). In agreement with previous studies the scores are summed to a total score ranging from 5 to 35. A score of 20 represents the midpoint between satisfied and dissatisfied with life.

SECONDARY OUTCOMES:
Disability Rating Scale (DRS) | through study completion, an average of one and a half months
  The Disability Rating Scale consists of eight items, each of which is rated on a scale of 0 to either 3 or 5.
Neurobehavioral Rating Scale-Revised (NBRS-R) | through study completion, an average of one and a half months
  The Neurobehavioral Rating Scale-revised (NBRS-R) is a widely-used measurement around the world, which focus specifically on brain injury patients. It appears to be a more sensitive tool for monitoring neurobehavioral disturbances. The NBRS-R consists of 29 items with a four-level response (absent, mild, moderate, severe).
Rancho Los Amigos Cognitive Scale-Revised (RLAS-R) | through study completion, an average of one and a half months
  Rancho Los Amigos Cognitive Scale-Revised (RLAS-R) was used to categorise level of cognitive and behavioral function. RLAS-R levels were dichotomised into 'inferior functioning' (RLAS-R 1-8) and 'superior functioning' (RLAS-R 9-10).
Functional Ambulation Classification Scale (FACS) | through study completion, an average of one and a half months
  The Functional Ambulation Classification Scale (FACS) classifies patients according to basic motor skills necessary for functional ambulation and ranges from independent walking outside (Category 5) to non-functional walking (Category 0)
Hospital Anxiety and Depression Scale | through study completion, an average of one and a half months
  Hospital Anxiety and Depression Scale is a scale which is a 14-item questionnaire. Seven items evaluate depression and the other seven items evaluate anxiety. Subscale total scores above 7 indicate an anxiety disorder or depression, respectively.
Pittsburgh Sleep Quality İndex (PSQI) | through study completion, an average of one and a half months
  The PSQI has 19 items assessing subjectively perceived sleep quality in the previous month. Global scores combine subdomains of sleep duration, sleep disturbance, sleep latency, sleep efficiency, daytime dysfunction, overall sleep quality and medication use. The score range is 0-21, with higher values indicating poorer sleep quality.
NHP (Nottingham Health Profile) | through study completion, an average of one and a half months
  The NHP is divided into two parts: part 1 comprises 38 statements divided into six domains (energy, pain, emotional reactions, sleep, social isolation, and physical mobility). Part 2 of the NHP, lists six important activities of daily living that are affected negatively if the patient has a poor state of health.

CONTACTS AND LOCATIONS:
Overall Officials: Fatma Özcan, MD, Principal Investigator — Gaziler Physical Medicine and Rehabilitation, Training and Research Hospital, Department of PMR
Locations (1):
- Fatma Özcan, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No